CLINICAL TRIAL: NCT00126386
Title: Zoledronic Acid (Zometa) for the Management of Tumor-induced Hypercalcemia (TIH) and Malignant Bone Pain (MBP) in the Community: A Feasibility Study
Brief Title: Zometa for the Management of Tumor-induced Hypercalcemia and Malignant Bone Pain in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17280; 17280
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-08

CONDITIONS: Cancer; Hypercalcemia; Pain
Keywords: tumor induced hypercalcemia; malignant bone pain; bisphosphonates; cancer; palliative; Zometa; palliative patient; treatment in community
MeSH Terms: conditions — Neoplasms; Hypercalcemia; Pain | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Zoledronic acid (Zometa)

SUMMARY:
Treatment in the home and hospice of long-term care facilities, particularly for non-ambulatory patients, could provide significant advantages for patients and for the region. The Calgary Health Region has a unique resource in the home parenteral therapy program (HPTP). With the assistance of HPTP, patients requiring bisphosphonate treatment for the management of tumor-induced hypercalcemia (TIH) or malignant bone pain (MBP) could be treated in the community (ie at home). However, the resources required and the costs associated with community-based (homes, hospices, long-term care facilities) treatment of TIH and MBP need to be identified and evaluated so as to guide future regional decision making.

DETAILED DESCRIPTION:
Treatment in the home and hospice of long-term care facilities, particularly for non-ambulatory patients, could provide significant advantages for patients and for the region. The Calgary Health Region has a unique resource in the home parenteral therapy program (HPTP). With the assistance of HPTP, patients requiring bisphosphonate treatment for the management of TIH or MBP could be treated in the community (ie at home). However, the resources required and the costs associated with community-based (homes, hospices, long-term care facilities) treatment of TIH and MBP need to be identified and evaluated so as to guide future regional decision making.

ELIGIBILITY:
Inclusion Criteria:

If hypercalcemic:

* Serum corrected Ca+++>= 2.5 mmol/L and symptomatic hypercalcemia
* Asymptomatic hypercalcemia with corrected Ca+++>= 3.0 mmol/L
* Moderate to severe intolerable pain (>=6/10 on numerical rating scale [NRS]) despite optimal treatments with a strong opioid such as morphine, hydromorphone, fentanyl, oxycodone or methadone
* Radiotherapy bone pain related to metastatic bone disease

Exclusion Criteria:

* Not on a regular bisphosphonate regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2004-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
feasibility of treating hypercalcemia in the community
resources required

CONTACTS AND LOCATIONS:
Overall Officials: Jose Pereira, MD, Principal Investigator — Alberta Cancerboard
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada